CLINICAL TRIAL: NCT02855840
Title: Qualitative Study of the Consequences of Auto-immune Diseases on Quality of Life
Brief Title: Auto-immune Diseases and Quality of Life
Acronym: QUALIMAIRAU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DEVILLIERS FMR 2014
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Systemic Auto-immune Diseases; Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (3):
- systemic lupus erythematous
  Interventions: Other: completion of the quality of life questionnaire
- systemic sclerosis
  Interventions: Other: completion of the quality of life questionnaire
- inflammatory myopathy
  Interventions: Other: completion of the quality of life questionnaire

INTERVENTIONS:
Other: completion of the quality of life questionnaire

SUMMARY:
Systemic lupus erythematous (SLE), systemic sclerosis (Ssc) and inflammatory myopathy (IM) are rare diseases, whose prevalence is estimated at 43, 15 and 10 cases, respectively, for 100 000 inhabitants in France. These diseases belong to the group of auto-immune diseases and require specialized follow-up in an expert centre. The repercussions of SLE, Ssc and IM on the everyday life of patients are heavy, and notably linked to skin involvement, to diminished functional capacities and psychological problems. The vast majority of these diseases concern middle-aged, professionally-active individuals, for whom the socio-professional repercussions are major and too often neglected. The aim of this study is to analyse the consequences of auto-immune diseases on quality of life. Current quality of life questionnaires are not suitable, and do not reveal the reality of the situation and its different nuances. In this research, the quality of life of patients will be envisaged through their everyday lives. How do these patients construct the social reality of the disease? How do they perceive their health status and their social situation? How do they organize their everyday lives around the disease: work, leisure, relationships with their entourage... ?

ELIGIBILITY:
Inclusion Criteria:

* For all patients:
* Patients aged 18 to 75 years
* Patients able to understand written and spoken French
* Patients who have been given oral and written information about the research

For patients with SLE:

- SLE defined by American College of Rheumatology (ACR) 1997 criteria

For patients with systemic sclerosis:

- SSc according to the Leroy or American Rheumatism Association (ARA) criteria

For patients with IM:

- IM according to the Trojanov criteria

Exclusion Criteria:

* Refusal to take part in the study
* Cognitive/psychological status incompatible with interviews

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Systemic lupus erythematous (SLE), systemic sclerosis (Ssc) and inflammatory myopathy (IM)
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
semi-directive individual interviews in the 3 groups of patients | day one

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France